CLINICAL TRIAL: NCT05813132
Title: BeEAM (Bendamustine, Etoposide, Cytarabine, Melphalan) Versus CEM (Carboplatin, Etoposide, Melphalan) in Lymphoma Patients as a Conditioning Regimen Before Autologous Hematopoietic Cell Transplantation
Brief Title: BeEAM Versus CEM in Lymphoma Patients as a Conditioning Regimen Before Autologous Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Associate Professor, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeEAM versus CEM in lymphoma
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — BEAM protocol; Bendamustine Hydrochloride; Etoposide; Cytarabine; Melphalan; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeEAM Regimen (Active Comparator): BeEAM (Bendamustine, Etoposide, Cytarabine, Melphalan)
  Interventions: Drug: BEAM Protocol
- CEM Regimen (Active Comparator): CEM (Carboplatin, Etoposide, Melphalan)
  Interventions: Drug: CEM protocol

INTERVENTIONS:
Drug: BEAM Protocol — BeEAM (Bendamustine, Etoposide, Cytarabine, Melphalan)
  Other Names: (Bendamustine, Etoposide, Cytarabine, Melphalan
  Arms: BeEAM Regimen
Drug: CEM protocol — CEM (Carboplatin, Etoposide, Melphalan)
  Other Names: (Carboplatin, Etoposide, Melphalan)
  Arms: CEM Regimen

SUMMARY:
The proposed research aims to compare between BeEAM standard regimen and CEM as conditioning regimen in lymphoma patients in safety profile& toxicity, infections (Febrile neutropenia) during transplant, time to engraftment (recovery not neutropenic), Length of stay at hospital, time to relapse, and other complications.

DETAILED DESCRIPTION:
1. All patients' history will be confirmed diagnosis of lymphoma subtype under microscope to When an abnormal cell called a Reed-Sternberg cell is present, the lymphoma is classified as Hodgkin if not so it is NHL Which has another subtype by phenotyping.
2. All patient will be confirmed in CR or PR before transplant was assessed by 18-FDG PET-CT imaging.
3. All patients will be mobilized by using G-CSF agent (filgrastim)

   * plerixafor
4. Check cluster of differentiation 34 (CD34+) count as Hematopoietic stem cell (HSCs) graft is mainly determined by the number of CD34+ cells present. the minimal number of CD34+ cells for an autologous transplant (Cutoff point) is <2 ×106 CD34+ cells/kg BW. Stem cell collection with target yield of 2-5 x 106 CD34 cells/kg (preferred) (13)
5. Collect HSCs from the patient prior to receipt of high-dose chemotherapy by Leukapheresis through central line on one or two sessions.
6. According to protocol of chemotherapy if BeEAM protocol, cells put in the final product includes 5-10% dimethyl sulfoxide (DMSO) as a cryoprotectant and 0.05-0.25" mL of ACD-A stabilizer solution per ml of transplant. Freezing at a controlled rate of 1-2"°C per minute if CME protocol cells will be mix with ACD and freezing (fresh cells).
7. All enrolled patients (50) will be randomly assigned into two equal arms:

   Arm A : will receive BeEAM regimen : Bendamustine on day
   * 7 and -6 dose of 160-200 mg/m2/day IV in a 2-h infusion, Etoposide 150-200 mg/m2/day BID infusion on 30 min with 500 ml NaCl 0.9% on days -5 to -2, cytarabine 200 mg/m2/d IV BID in a 30-min infusion with 500 ml NaCl 0.9% on days -5 to -2, and melphalan 140 mg/m2 IV in a single 1-h 500 ml infusion with 0.9% NaCl on day -1(12)

   Arm B: will receive CME regimen: Carboplatin 25m/kg for day-2 and -1 in a 1hr infusion, Melphalan 140mg/m2 for day-2 and -1 in a 30 min infusion, Etoposide 30m/kg for day-2 and -1 in 2-3 hr.
8. All patients received granulocyte - colony stimulating factor (G-CSF) at 5 ug/kg BW. starting from day +4 after AHSCT until absolute neutrophil count reached 1.5 × 109/l for two consecutive days. All patients received antiviral (oral acyclovir), antifungal (Oral fluconazole), and antibacterial (oral levofloxacin) prophylaxis. Since the start of conditioning until patient not neutropenic (Count reached 0.5 × 109/l), hyperuricemia prophylaxis was given (Oral allopurinol 100 mg TID), hepatic veno-occlusive disease prophylaxis enoxaparin sc daily until platelet > 25000/mm3 and ursodeoxycholic acid.

   transfusion of platelets or red blood cells was given when platelet count was lower than 20 × 109/l or hemoglobin level was lower than 80 g/l, respectively.
9. Monitoring for any possible side effects:
10. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.

ELIGIBILITY:
Inclusion Criteria

1. Patients with lymphoma relapsed/refractory (RR) Hodgkin's lymphoma (HL) and non-Hodgkin lymphoma (NHL) with all subtypes. 2. Treat with conventional dose salvage regimens 3. Remission status before HSCT is complete remission (CR) or partial remission (PR).

4. Age>18 years. 5. Gender male and female. 6. CD34+ count cells <2 ×106 CD34+ cells/kg BW. Exclusion Criteria

1. Remission status before HSCT is non remission (NR) or progressive disease (PD).
2. CD34+ count cells <2 ×106 CD34+ cells/kg BW
3. CNS lymphoma or solid tumor not included in population.
4. Pregnancy or breast-feeding.
5. Any Psychological, familial, sociological, or geographical factor that interfere with patient adherence to medications.
6. History of allergy to any medications in both protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Side Effects. | 3 month
  Side effects of treatment

SECONDARY OUTCOMES:
Concentration of CD34+ | Three Months
  CD34+

CONTACTS AND LOCATIONS:
Overall Officials: Noha A. El bassiouny, Lecturer, Study Director — Damanhour University; Mohamed Khalef, Ph.D, Study Director — Maady Military Hospital; Mahmoud Abdallah, Ph.D., Study Director — International Medical Center (IMC) Hospital, Cairo, Egypt.
Locations (1):
- International Medical Center (IMC) Hospital, Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Velasquez WS, Cabanillas F, Salvador P, McLaughlin P, Fridrik M, Tucker S, Jagannath S, Hagemeister FB, Redman JR, Swan F, et al. Effective salvage therapy for lymphoma with cisplatin in combination with high-dose Ara-C and dexamethasone (DHAP). Blood. 1988 Jan;71(1):117-22. PMID 3334893
- [Result] Frankiewicz A, Sadus-Wojciechowska M, Najda J, Czerw T, Mendrek W, Sobczyk-Kruszelnicka M, Soska K, Ociepa M, Holowiecki J, Giebel S. Comparable safety profile of BeEAM (bendamustine, etoposide, cytarabine, melphalan) and BEAM (carmustine, etoposide, cytarabine, melphalan) as conditioning before autologous haematopoietic cell transplantation. Contemp Oncol (Pozn). 2018;22(2):113-117. doi: 10.5114/wo.2018.77046. Epub 2018 Jun 30. PMID 30150889
- [Derived] Eltelbanei MA, El-Bassiouny NA, Abdalla MS, Khalaf M, Werida RH. Clinical and safety outcomes of BeEAM (Bendamustine, Etoposide, Cytarabine, Melphalan) versus CEM (Carboplatin, Etoposide, Melphalan) in lymphoma patients as a conditioning regimen before autologous hematopoietic cell transplantation. BMC Cancer. 2024 Aug 13;24(1):1002. doi: 10.1186/s12885-024-12694-9. PMID 39134959